CLINICAL TRIAL: NCT05128123
Title: Influence of Social Determinants of Health on the Management of Hepatocellular Carcinoma in the French National Cohort Study CHIEF
Brief Title: Influence of Social Determinants of Health on the Management of HCC in the French National Cohort Study CHIEF
Acronym: SOCIAL-CHIEF
Status: Active, not recruiting | Type: Observational
Sponsor: University Hospital, Grenoble (Other)
Collaborators: University Grenoble Alps (Other); University Hospital, Caen (Other); Amiens University Hospital (Other); National Cancer Institute, France (Other Government)
Responsible Party: Sponsor
Other Study IDs: 38RC21.0295
Record Dates: First submitted 2021-10-28; First posted 2021-11-19 (Actual); Last update posted 2025-04-20 (Actual); Status verified 2025-04

CONDITIONS: Hepatocellular Carcinoma
Keywords: Hepatocellular Carcinoma; Primary Liver Cancer; Social determinants of health
MeSH Terms: conditions — Carcinoma, Hepatocellular

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
With 8,000 related deaths per year, HCC is one of the most dangerous cancers in France. The main reason for the poor prognosis of HCC is most often a diagnosis at an advanced stage ineligible for curative treatment. In the field of oncology, low participation to screening is closely linked to socioeconomic status (e.g. level of education, income, employment). In HCC, the socioeconomic status is linked to incidence, overall survival and treatment allocation in US, UK and Australia. This suggests that the social environment should be taken into account when designing interventions and policies that allows facilitating the medical pathways for patients with HCC with the ultimate goal of improving the overall prognosis. However, the studies assessing the impact of social determinants on the management of HCC in France are limited. Bryère at al. reported that the highest incidence and the worst prognosis of HCC were observed in the most disadvantaged populations in France. To date, there is no available data concerning the influence of social determinants on: implementation of surveillance programs of HCC, stage of disease at the time of diagnosis or treatment allocation. This data is essential for better understanding the geographic disparities observed in France and for developing the strategies to remedy them.

CHIEF is a multicenter longitudinal observational study of patients with HCC (ClinicalTrials.gov Identifier: NCT04348838), that will collect the exhaustive data including patient and tumor characteristics, diagnostic circumstances and modalities, care pathway from diagnostic imaging to referral to expert center, treatment allocation and implementation, and 5-year follow up including recurrent assessment of quality of life.

Social-CHIEF is an ancillary study to the CHIEF cohort (approved by CHIEF scientific committee). The population of this study will consist in a subset of patients from the CHIEF prospectively included or already recruited who accept to participate in this study. The data collected in CHIEF will be retrieved from the CHIEF main database and additional data about social determinants will be specifically investigated by self-administrated questionnaires. The results obtained will provide a better understanding of the influence of social determinants on health trajectories of HCC patients. These data will be essential in recommending new health policies and in designing innovative intervention studies to address social disparities.

ELIGIBILITY:
Inclusion Criteria:

* Patients already included in the French national CHIEF cohort who accept to participate in the Social-CHIEF study.

Exclusion Criteria:

* Patients included in CHIEF cohort who opposed to participate in the Social-CHIEF study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients (18 years old and older) with newly diagnosed or already known HCC that are eligible for systemic treatments and already included in the national CHIEF cohort.
Sampling Method: Non-Probability Sample
Enrollment: 1600 (Estimated)
Dates: Start 2022-01-21 (Actual); Primary Completion 2024-12-31 (Actual); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
The primary objective will be to assess the rates of curative treatment (either resection, ablation or liver transplantation) according to the social determinants of health | Up to 3 months
  Treatment allocation will be retrieved from the CHIEF eCRF and categorized into curative treatment (either ablation, resection or liver transplant) or non-curative treatments (all other treatment options). Rates of curative treatments will be described across categories of the different social determinants of health. Crude and adjusted relative risks between these determinants and the primary outcome will be estimated using a generalized linear regression model.

SECONDARY OUTCOMES:
Describe the underlying etiology, clinical and biological characteristics of HCC, diagnostic modalities, therapeutic management according to social determinants of health | Up to 3 months
  Descriptive analysis of the underlying etiology, patient characteristics and tumor stage at the time of diagnosis, diagnostic methods (as part of the surveillance program vs. incidental), therapeutic management (curative vs. non-curative) and distribution of the different treatment modalities (transplantation, resection, percutaneous destruction, chemoembolization, intra-arterial radiotherapy, systemic treatments), compliance with management recommendations and care pathways, according to indicators of social determinants of health.
Assessment of the relationship between social health determinants and one-year survival | Up to 3 months
  Progression-free survival (PFS) and overall survival (OS) parameters that will be retrieved from the CHIEF eCRF. The determinants of PFS and OS at one-year will be assessed using a survival model.
Assessment of the relationship between social health determinants and quality indicators for the management of HCC (diagnosis at 2 years after treatment) | Up to 3 months
  The quality indicators for the management of HCC will be retrieved from the CHIEF eCRF. The determinants of the quality indicators for the management of HCC (from diagnosis to 2 years after treatment) will be evaluated using a logistic regression model.
Assessment of the relationship between social health determinants and the quality of life of patients at 6 and 18 months after inclusion in the CHIEF cohort study | Up to 3 months
  The quality of life of patients is assessed using the EQ-5D-5L questionnaire, the QLQ-C30 questionnaire and its module HCC18 specific to the HCC at different time points (6 months and 18 months from inclusion) during the follow-up in the CHIEF cohort. The determinants of a degraded quality of life will be evaluated using logistic regression.

CONTACTS AND LOCATIONS:
Overall Officials: Charlotte E Costentin, Pr, Principal Investigator — University Hospital, Grenoble
Locations (1):
- Anna M Borowik, La Tronche, Auvergne-Rhône-Alpes, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Costentin CE, Mourad A, Lahmek P, Causse X, Pariente A, Hagege H, Dobrin AS, Becker C, Marks B, Bader R, Condat B, Heluwaert F, Seitz JF, Lesgourgues B, Denis J, Deuffic-Burban S, Rosa I, Decaens T; CHANGH Study Group. Hepatocellular carcinoma is diagnosed at a later stage in alcoholic patients: Results of a prospective, nationwide study. Cancer. 2018 May 1;124(9):1964-1972. doi: 10.1002/cncr.31215. Epub 2018 Mar 28. PMID 29589878
- [Background] Damiani G, Basso D, Acampora A, Bianchi CB, Silvestrini G, Frisicale EM, Sassi F, Ricciardi W. The impact of level of education on adherence to breast and cervical cancer screening: Evidence from a systematic review and meta-analysis. Prev Med. 2015 Dec;81:281-9. doi: 10.1016/j.ypmed.2015.09.011. Epub 2015 Sep 25. PMID 26408405
- [Background] Herbert C, Launoy G, Gignoux M. Factors affecting compliance with colorectal cancer screening in France: differences between intention to participate and actual participation. Eur J Cancer Prev. 1997 Feb;6(1):44-52. doi: 10.1097/00008469-199702000-00008. PMID 9161812
- [Background] Jembere N, Campitelli MA, Sherman M, Feld JJ, Lou W, Peacock S, Yoshida E, Krahn MD, Earle C, Thein HH. Influence of socioeconomic status on survival of hepatocellular carcinoma in the Ontario population; a population-based study, 1990-2009. PLoS One. 2012;7(7):e40917. doi: 10.1371/journal.pone.0040917. Epub 2012 Jul 13. PMID 22808283
- [Background] Singal AG, Li X, Tiro J, Kandunoori P, Adams-Huet B, Nehra MS, Yopp A. Racial, social, and clinical determinants of hepatocellular carcinoma surveillance. Am J Med. 2015 Jan;128(1):90.e1-7. doi: 10.1016/j.amjmed.2014.07.027. Epub 2014 Aug 10. PMID 25116425
- [Background] Clark PJ, Stuart KA, Leggett BA, Crawford DH, Boyd P, Fawcett J, Whiteman DC, Baade PD. Remoteness, race and social disadvantage: disparities in hepatocellular carcinoma incidence and survival in Queensland, Australia. Liver Int. 2015 Dec;35(12):2584-94. doi: 10.1111/liv.12853. Epub 2015 May 22. PMID 25900432
- [Background] Bryere J, Dejardin O, Bouvier V, Colonna M, Guizard AV, Troussard X, Pornet C, Galateau-Salle F, Bara S, Launay L, Guittet L, Launoy G. Socioeconomic environment and cancer incidence: a French population-based study in Normandy. BMC Cancer. 2014 Feb 13;14:87. doi: 10.1186/1471-2407-14-87. PMID 24524213
- [Background] Tron L, Belot A, Fauvernier M, Remontet L, Bossard N, Launay L, Bryere J, Monnereau A, Dejardin O, Launoy G; French Network of Cancer Registries (FRANCIM). Socioeconomic environment and disparities in cancer survival for 19 solid tumor sites: An analysis of the French Network of Cancer Registries (FRANCIM) data. Int J Cancer. 2019 Mar 15;144(6):1262-1274. doi: 10.1002/ijc.31951. Epub 2018 Dec 3. PMID 30367459
- See also: INSERM CépiDc - Causes of death from 1979 to 2014 — http://cepidc-data.inserm.fr/inserm/html/index2.htm